CLINICAL TRIAL: NCT02537561
Title: A Phase I Adaptive Design Trial of Talazoparib in Combination With Gemcitabine and Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Talazoparib in Combination With Gemcitabine and Cisplatin in Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The pharmaceutical company did not want to follow through with support for the study.
Sponsor: Washington University School of Medicine (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-x279
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Solid Tumors; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Cisplatin, Gemcitabine, Talazoparib Solid Tumors (Experimental): * Dose levels of the drugs will be dependent on which dose level the participants is enrolled.
  * Cisplatin will be infused as a 30 minute intravenous piggyback (IVPB) on Day 1 of each 21 day cycle.
  * Gemcitabine will be infused as a 30 minute IVPB on Days 1 and 8 of each 21 day cycle. On day 1, gemcitabine will be given before cisplatin.
  * Talazoparib will be started with cycle 2. It is an oral drug which will be administered on an outpatient basis daily.
  * Cisplatin and gemcitabine will be given for a total of 6 cycles.
  * Talazoparib may be continued as a single agent maintenance therapy.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Talazoparib
- Arm 2: Cisplatin, Gemcitabine, Talazoparib NSCLC (Experimental): * Dose levels of the drugs will depend on what the MTD is in the dose escalation portion of the study
  * Cisplatin will be infused as a 30 minute intravenous piggyback (IVPB) on Day 1 of each 21 day cycle.
  * Gemcitabine will be infused as a 30 minute IVPB on Days 1 and 8 of each 21 day cycle. On day 1, gemcitabine will be given before cisplatin.
  * Talazoparib will be started with cycle 2. It is an oral drug which will be administered on an outpatient basis daily.
  * Cisplatin and gemcitabine will be given for a total of 6 cycles.
  * Talazoparib may be continued as a single agent maintenance therapy.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Talazoparib

INTERVENTIONS:
Drug: Cisplatin
  Other Names: cis-DDP; cis-Platinum II; cis-Diamminedichloroplatinum; DDP
Drug: Gemcitabine
  Other Names: Gemzar®
Drug: Talazoparib
  Other Names: BMN 673

SUMMARY:
In this proposed study the investigators will combine gemcitabine and cisplatin with talazoparib to determine the recommended Phase 2 dose (RP2D) of this combination regimen. After determination of the RP2D patients with lung cancer whose tumors carry molecular alterations in DNA repair pathway genes will be enrolled to an expansion cohort to determine anti-tumor efficacy. Tissue samples of patients with confirmed partial response, complete response, and non-responders will be obtained for whole exome, and transcriptome sequencing to characterize the genetic alterations associated with response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced solid tumor for which no curative standard treatment options exist and for which gemcitabine and cisplatin is a suitable treatment regimen.
* After the determination of the maximum tolerated dose, an expansion cohort of 20 patients with non-small cell lung cancer whose tumors demonstrate variants in DNA repair pathway genes will be enrolled.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Prior treatment for this disease is allowed if it has been completed at least 2 weeks prior to study enrollment and if all treatment-related toxicities are resolved. Prior exposure to a PARP inhibitor is allowed for patients in the dose-finding portion of the study.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
  * Tissue available for sequencing (either archival tissue or readily accessible tumor for fresh routine biopsy).
  * Able to swallow tablets.
  * Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
  * Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Received any other investigational agent within 2 weeks of starting the first dose on study.
* Symptomatic brain metastases. Known brain metastases are allowed if asymptomatic and previously treated. Patients must be at least 4 weeks post-brain radiation therapy.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, gemcitabine, talazoparib, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active coronary artery disease, uncontrolled seizure, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Safety and toxicities as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 30 days after completion of treatment (estimated average to be 7 months)
Maximum tolerated dose (MTD) | Completion of dose escalation portion of study (approximately 12 months)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 30% of patients in a cohort are expected to experience a dose-limiting toxicity (DLT) during the second cycle based on the CRM algorithm. Dose escalations will proceed until the MTD is determined.
Objective response rate (ORR) in preselected patients with BRCAness tumoral genotype | Up to completion of treatment (estimated average of 6 months)
  ORR - proportion of patients who achieved a complete response or a partial response

SECONDARY OUTCOMES:
Disease control rate (DCR) | Until death (estimated average to be 12 months)
  * DCR - percentage of participants who have achieved complete response, partial response, and stable disease
  * Complete response: disappearance of all lesions and normalization of tumor marker level
  * Partial response: at least a 30% decrease in the sum of the diameters of target lesions and no new lesions
  * Stable disease: neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease
Progression-free survival (PFS) | Until death (estimated average to be 12 months)
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  -Progressive disease - At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one more new lesions PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Objective response rate (ORR) | Up to completion of treatment (estimated average of 6 months)
  ORR - proportion of patients who achieved a complete response or a partial response
Overall survival (OS) | Until death (estimated average to be 12 months)
  OS: duration of time from start of treatment to time of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Saiama Waqar, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu